CLINICAL TRIAL: NCT01275339
Title: Aortic Stenosis and PhosphodiEsterase Type 5 iNhibition (ASPEN): A Pilot Study
Acronym: ASPEN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty enrolling patients and PI moved institutions.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-1334b
Record Dates: First submitted 2011-01-06; First posted 2011-01-12 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Aortic Stenosis; LV Remodeling, Hypertrophy
Keywords: Aortic valve stenosis; Tadalafil; Phosphodiesterase inhibitors; Hypertension, pulmonary; Hypertrophy, left ventricular
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertrophy; Hypertension, Pulmonary; Hypertrophy, Left Ventricular | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tadalafil in Diabetic Cohort (Active Comparator)
  Interventions: Drug: Tadalafil
- Placebo in Diabetic Cohort (Placebo Comparator)
  Interventions: Drug: Placebo
- Tadalafil in Non-Diabetic Cohort (Active Comparator)
  Interventions: Drug: Tadalafil
- Placebo in Non-Diabetic Cohort (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Active drug will be encapsulated to look identical to the placebo pill. Subjects will take a single oral dose of tadalafil once daily from the time of randomization until study completion (6 months). Subjects will begin by taking 20 mg (1 pill) daily for 3 days before having the dose increased to 40 mg (2 pills) once daily. If the increase to 40mg daily is not tolerated, then the dose will be decreased back to 20mg daily.
  Other Names: Cialis; Adcirca
  Arms: Tadalafil in Diabetic Cohort; Tadalafil in Non-Diabetic Cohort
Drug: Placebo — The placebo pill will be encapsulated to look identical to the active drug pill. Subjects will take a single oral dose of placebo once daily from the time of randomization until study completion (6 months). Subjects will begin by taking 1 pill daily for 3 days before having the dose increased to 2 pills once daily. If the increase to 2 pills is not tolerated, then the dose will be decreased back to 1 pill daily.
  Arms: Placebo in Diabetic Cohort; Placebo in Non-Diabetic Cohort

SUMMARY:
Currently, aortic stenosis (AS) is considered a "surgical disease" with no medical therapy available to improve any clinical outcomes, including symptoms, time to surgery, or long-term survival. Thus far, randomized studies involving statins have not been promising with respect to slowing progressive valve stenosis. Beyond the valve, two common consequences of aortic stenosis are hypertrophic remodeling of the left ventricle (LV) and pulmonary venous hypertension; each of these has been associated with worse heart failure symptoms, increased operative mortality, and worse long-term outcomes. Whether altering LV structural abnormalities, improving LV function, and/or reducing pulmonary artery pressures with medical therapy would improve clinical outcomes in patients with AS has not been tested. Animal models of pressure overload have demonstrated that phosphodiesterase type 5 (PDE5) inhibition influences nitric oxide (NO) - cyclic guanosine monophosphate (cGMP) signaling in the LV and favorably impacts LV structure and function, but this has not been tested in humans with AS. Studies in humans with left-sided heart failure and pulmonary venous hypertension have shown that PDE5 inhibition improves functional capacity and quality of life, but patients with AS were not included in those studies. The investigators hypothesize that PDE5 inhibition with tadalafil will have a favorable impact on LV structure and function as well as pulmonary artery pressures. In this pilot study, the investigators anticipate that short-term administration of tadalafil to patients with AS will be safe and well-tolerated.

DETAILED DESCRIPTION:
Subjects with moderately severe to severe aortic stenosis (AS), left ventricular hypertrophy (LVH), diastolic dysfunction, preserved ejection fraction, and no planned aortic valve replacement over the next 6 months will be eligible for this randomized, double-blind, placebo-controlled, pilot study. There will be a diabetic cohort (n=32) and non-diabetic cohort (n=24); each cohort will be randomized 1:1 to tadalafil vs. placebo. During a baseline study visit, the following will be obtained: clinical data, 6 minute walk, quality of life questionnaire, blood draw, and an echocardiogram. A 3-day run-in will occur to initially assess tolerability and compliance. If the drug is tolerated during this run-in period, participants will be randomized. An MRI will also be performed during this randomization visit. Follow-up study visits and testing will occur at 6 and 12 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe aortic stenosis (AVA < 1.5 cm2)
* Left ventricular hypertrophy
* Diastolic dysfunction as evidenced by tissue Doppler e' (average of septal and lateral) ≤ 7 cm/s
* EF ≥ 50%
* None or minimal symptoms related to aortic stenosis (NYHA ≤ 2)
* The subject and treating physician are not planning on a valve replacement procedure to occur during the next 6 months
* Ambulatory
* Normal sinus rhythm
* 18 years of age and older
* Able and willing to comply with all the requirements for the study

Exclusion Criteria:

* Need for ongoing nitrate medications
* SBP < 110mmHg or MAP < 75mmHg
* Moderately severe or severe mitral regurgitation
* Moderately severe or severe aortic regurgitation
* Contraindication to MRI
* Creatinine clearance < 30 mL/min
* Cirrhosis
* Pulmonary fibrosis
* Increased risk of priapism
* Retinal or optic nerve problems or unexplained visual disturbance
* If a subject requires ongoing use of an alpha antagonist typically used for benign prostatic hyperplasia (BPH) (prazosin, terazosin, doxazosin, or tamsulosin), SBP < 120 mmHg or MAP < 80 mmHg is excluded
* Need for ongoing use of a potent CYP3A inhibitor or inducer (ritonavir, ketoconazole, itraconazole, rifampin)
* Current or recent (≤ 30 days) acute coronary syndrome
* O2 sat < 90% on room air
* Females that are pregnant or believe they may be pregnant
* Any condition which the PI determines will place the subject at increased risk or is likely to yield unreliable data
* Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian R. Lindman, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tadalafil in Diabetic Cohort | Placebo in Diabetic Cohort | Tadalafil in Non-Diabetic Cohort | Placebo in Non-Diabetic Cohort
Started | 2 | 0 | 4 | 4
Completed | 1 | 0 | 3 | 4
Not Completed | 1 | 0 | 1 | 0
Not completed — Referred for surgery for AS symptoms | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were a small number of subjects enrolled in this trial before it was terminated. There was block randomization and none got assigned to the Diabetic placebo cohort. Only 2 diabetics were enrolled and they were both randomized to tadalafil.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil in Diabetic Cohort | Placebo in Diabetic Cohort | Tadalafil in Non-Diabetic Cohort | Placebo in Non-Diabetic Cohort | Total
Number analyzed (Participants) | 2 | 0 | 4 | 4 | 10
Age, Continuous [Mean (Full Range); unit: years] | 65 [62 to 68] |  | 81.25 [62 to 92] | 75.5 [59 to 89] | 75.7 [59 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2
  Male | 2 | 0 | 3 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0 | 0
  Asian | 0 |  | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0 | 0
  Black or African American | 1 |  | 1 | 0 | 2
  White | 1 |  | 3 | 4 | 8
  More than one race | 0 |  | 0 | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Diastolic Function as Measured by Tissue Doppler e'
Description: Measurement of e' (average of septal and lateral) on echo at each of the time points specified.
Time Frame: Baseline, 12 weeks, and 6 months
Population: There were 0 enrolled that were randomized to placebo in the diabetic cohort; the total number enrolled in the study was small, so this happened randomly.
Measure: Mean (Full Range); unit: cm/sec
Arm/Group | Tadalafil in Diabetic Cohort | Placebo in Diabetic Cohort | Tadalafil in Non-Diabetic Cohort | Placebo in Non-Diabetic Cohort
Number analyzed (Participants) | 2 | 0 | 4 | 4
cm/sec
  Baseline | 4.59 [3.52 to 5.65] |  | 5.97 [5.00 to 6.52] | 5.28 [4.48 to 6.21]
  12 weeks | 3.75 [3.21 to 4.28] |  | 6.44 [5.31 to 7.21] | 4.88 [4.36 to 5.61]
  6 months | 4.63 [3.91 to 5.34] |  | 6.16 [4.77 to 7.03] | 5.33 [3.57 to 6.18]

2. Secondary Outcome: Change in Myocardial Fibrosis (ECV) on MRI
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in Other Echocardiographic Indices of Diastolic Function
Description: E/e' and deceleration time
Time Frame: 12 weeks and 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Safety and Tolerability
Description: The following with be reported - frequency of the following: hypotension (SBP < 90 mmHg), symptomatic hypotension (symptoms of presyncope or syncope associated with SBP <90), syncope, hospitalization for a cardiac reason, myocardial infarction, new onset or worsening heart failure, and new sustained arrhythmia requiring intervention
Time Frame: 6 and 12 weeks and 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Indices of Systolic Function
Description: Stroke volume, EF, LV twist, and stress-corrected midwall shortening by echo and 3D multiparametric strain and EF by MRI
Time Frame: 12 weeks and 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in LV Hypertrophic Remodeling
Description: Relative wall thickness, LV chamber dimensions, and wall thickness
Time Frame: 12 weeks and 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Novel Echocardiographic Indices of Diastolic Function
Description: LV stiffness, viscoelasticity, and a load independent index of diastolic filling
Time Frame: 12 weeks and 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Change in 6 Minute Walk Distance
Time Frame: 6 and 12 weeks and 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in Circulating Neurohormonal Markers
Description: BNP and systemic markers of collagen turnover and oxidative stress
Time Frame: 6 and 12 weeks and 6 months
Reporting Status: Not Posted

10. Secondary Outcome: Change in Quality of Life
Description: Assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Time Frame: 6 and 12 weeks and 6 months
Reporting Status: Not Posted

11. Secondary Outcome: Change in Pulmonary Artery Pressure and Pulmonary Vascular Resistance as Assessed by Echo
Time Frame: 12 weeks and 6 months
Reporting Status: Not Posted

12. Secondary Outcome: Change in Systemic Blood Pressure
Time Frame: 6 and 12 weeks and 6 months
Reporting Status: Not Posted

13. Secondary Outcome: Change in RV Function
Description: TAPSE, s' tissue Doppler, and Tei index
Time Frame: 12 weeks and 6 months
Reporting Status: Not Posted

14. Secondary Outcome: Change in AS Severity
Description: Aortic valve area, transvalvular pressure gradients
Time Frame: 12 weeks and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: In that arm of the study, no patients were enrolled.
Arm/Group | Tadalafil in Diabetic Cohort | Placebo in Diabetic Cohort | Tadalafil in Non-Diabetic Cohort | Placebo in Non-Diabetic Cohort
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0 | 2/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil in Diabetic Cohort (N=2) | Placebo in Diabetic Cohort (N=0) | Tadalafil in Non-Diabetic Cohort (N=4) | Placebo in Non-Diabetic Cohort (N=4)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0 (0) | 1 (1) — Shortness of breath developed during the intervention period
orthopnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0 (0) | 0 (0) — Occurred during follow-up
lightheadedness (Cardiac disorders) | 1 (1) | NA | 0 (0) | 0 (0) — Occurred during follow-up
fall (Musculoskeletal and connective tissue disorders) | 0 (0) | NA | 1 (1) | 0 (0) — Unrelated to study drug as blood pressure was fine beforehand
dilated aorta (Vascular disorders) | 0 (0) | NA | 0 (0) | 1 (1) — Identified in follow-up although it may have been present at baseline
unsteady (Musculoskeletal and connective tissue disorders) | 0 (0) | NA | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | NA | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT01275339/Prot_SAP_000.pdf